CLINICAL TRIAL: NCT04356326
Title: Chronic Hypertension and Acetyl Salicylic Acid in Pregnancy, a Multicenter Prospective Randomized Double-blind Placebo-controlled Trial.
Brief Title: Chronic Hypertension and Acetyl Salicylic Acid in Pregnancy
Acronym: CHASAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHASAP; 2018-004160-58 (EudraCT Number)
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hypertension Complicating Pregnancy; Pre-Eclampsia; Intrauterine Growth Restriction; Aspirin; Perinatal Death; Placental Abruption
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Perinatal Death; Abruptio Placentae | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Prospective multicentric randomized double-blind superiority trial, placebo-controlled, on two parallel arms
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treatment will be administered double blind. Pouches or tablets and caskets will be indistinguishable, prepared in advance and made available to pharmacies in participating hospitals by the sponsor. The treatment boxes are given as the monthly visits to the patient, a reassignment box will be required on the server at each visit to obtain a new cabinet number. The cabinet number (detachable label) used at each visit will be reported in the patient's file.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin 150 mg (Experimental): Aspirin 150 mg / day (acetylsalicylic acid) once daily in the evening
  Interventions: Drug: Aspirin 150 mg
- Placebo (Placebo Comparator): Placebo taken in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 150 mg — Treatment assigned by randomization will be prescribed immediately and continued throughout pregnancy up to 35 weeks + 6 days for both groups. The active or placebo will be dispensed by the centre's pharmacy. Treatment will be taken in the evening. A daily log is given to patients and must be completed every day.
  Other Names: Active arm
  Arms: Aspirin 150 mg
Drug: Placebo — Treatment assigned by randomization will be prescribed immediately and continued throughout pregnancy up to 35 weeks + 6 days for both groups. The active or placebo will be dispensed by the centre's pharmacy. Treatment will be taken in the evening. A daily log is given to patients and must be completed every day.
  Other Names: comparator arm
  Arms: Placebo

SUMMARY:
A randomized clinical trial to assess the efficiency of acetylsalicylic acid (aspirin) 150 mg/day started before 20 weeks of gestation in the prevention on maternal and fœtal complications in pregnant women with chronic hypertension.

DETAILED DESCRIPTION:
Chronic hypertension affects 1 to 5% of women of childbearing age. According to the literature, about 45% of pregnant women with chronic hypertension will develop complications such as superimposed preeclampsia (PE), placental abruption, Intra Uterine Growth Restriction (IUGR), perinatal death, maternal death, or preterm delivery. To date, there is no curative treatment of vascular complications of chronic hypertension during pregnancy. The only effective treatment, once the complications are established, is usually stopping the pregnancy and delivering the placenta. The preventive treatment of these complications is therefore an important axis in the improvement of maternal and perinatal health.

Due to the very high risk of superimposed PE in chronic hypertensive patients and despite the lack of objective evidence of the effectiveness of low-dose aspirin in the prevention of superimposed PE in this population, the NICE (National Institute for Health and Care Excellence), associated with the Royal College of Gynecology-Obstetrics, recommends since 2010-2011 the use of low-dose aspirin in the prevention of this complication in chronic hypertensive pregnant women; then it was followed by the "U.S. Preventive Services Task Force (USPTF)" in 2014. Recently, the American College of Obstetrics and Gynecology (ACOG) adopted the suggestions of the USPTF and issued the same recommendations in 2018. The French college of obstetric (CNGOF: National College of French Gynecologists and Obstetricians), however, does not recommend the use of low-dose aspirin in pregnant chronic hypertensive women because of insufficient data.

Indeed, although the efficacy of low-dose aspirin is assumed in patients with previous PE, few studies have evaluated its efficacy in patients with chronic hypertension. Moreover, most of the controlled prospective studies using very low doses of aspirin (less than 100 mg) and starting after 20 weeks of gestation do not seem conclusive. For these reasons, the investigators propose to conduct a prospective randomized double-blind placebo-controlled trial to analyze the effectiveness of aspirin dosed at 150 mg and introduced before 20 weeks of gestation in women with chronic hypertension.

The primary endpoint is a maternal and perinatal composite morbidity and mortality including superimposed PE, intrauterine growth restriction, preterm delivery < 37 weeks of gestation, placental abruption, perinatal death, or maternal death.

The definition of superimposed PE in our study is the appearance of significant proteinuria in a chronic hypertensive pregnant woman.

In a secondary analyze, the statistician will use the new definition of superimposed PE that does not require the mandatory presence of proteinuria but the association of chronic hypertension and the appearance of neurological signs (eclampsia, persistent headache, visual disturbances, severe nausea or vomiting), pulmonary edema, persistent epigastric pain, thrombocytopenia <100000 platelets/µL, liver enzymes at 2 times normal, renal insufficiency ( serum creatinine ≥ 97 μmol/L or 1.1 mg/dL,) or a doubling of serum creatinine in the absence of chronic renal disease or significant proteinuria after 20 weeks of gestation or postpartum.

Significant proteinuria is defined as greater than 300 mg/24 hours or when the ratio proteinuria/ creatininuria is ≥ 30 mg/mmol (ratio to 0.3 if all are in mg/dL), in a non-proteinuric women with no urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient between 10 and 19 weeks of gestation + 6 days
* Chronic hypertension, whether treated or not, know before pregnancy or diagnosed before randomization
* Singleton pregnancy
* Signed the written informed consent
* Affiliation to social security

Exclusion Criteria:

* ---Medical history requiring anticoagulation (antiphospholipid syndrome, deep vein thromboembolic disease, pulmonary embolism, atherothrombosis, patient with mechanical heart valves),
* Patient receiving aspirin for another indication outside pregnancy,
* Patient with significant proteinuria (> 300mg/24 hours or a proteinuria/creatininuria ratio ≥ 30mg/mmol),
* Active bleeding,
* History of severe PE with delivery < 34 weeks of gestation,
* Hypersensitivity to salicylates such as aspirin and other nonsteroidal anti-inflammatory drugs (NSAIDs),
* Platelet count lower than 100,000 cells/microliter (dosage less than 6 months old),
* Hemostasis disorders, including hemophilia (with thrombocytopenia)
* Any constitutional or acquired hemorrhagic disease, (including digestive hemorrhages, history of hemorrhagic stroke and thrombocytopenia
* Human immunodeficiency virus, or hepatitis B virus, or hepatitis C virus positive serum,
* Patient included in another interventional study which could interfere with the results of the study,
* Age <18 years old,
* Women under the protection of justice,
* Patients with psychiatric follow-up, poor understanding of French or cognitive problems,
* Duodenal ulcer,
* Severe renal impairment,
* Severe hepatic insufficiency,
* Severe cardiac impairment,
* Gout,
* Patients with known glucose-6-phosphate dehydrogenase deficiency,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Composite morbidity-mortality criterion including preeclampsia, intra-uterine growth retardation <10th percentile, placental abruption, Preterm birth < 37 weeks of gestation, Perinatal death, Maternal death | 9 months
  A composite morbidity-mortality criterion that includes the occurrence during pregnancy or postpartum of at least one of the following events: preeclampsia, IUGR <10th percentile, placental abruption, Preterm birth < 37 weeks of gestation, Perinatal death (death from 22 weeks of gestation until 28 days after birth), Maternal death

SECONDARY OUTCOMES:
IUGR (< 10th percentile of birth weight) | 9 months
  Rate of IUGR (< 10th percentile of birth weight)
Placental abruption | 9 months
  Rate of placental abruption
Preterm birth < 37 weeks of gestation | 9 months
  Rate of severe preterm delivery (< 37 weeks of gestation)
Maternal death | 9 months
  Rate of severe maternal death
Severe pre-eclampsia | 9 months
  Rate of severe pre-eclampsia. Concerning the rate of superimposed PE, it will be analyze according the two definition specified in the rational
Intrauterine growth restriction (IUGR) | 9 months
  Rate of severe IUGR (< 5th percentile of birth weight)
Preterm delivery | 8 months
  Rate of severe preterm delivery (< 34 weeks of gestation)
Fetal loss | 5 months
  Rate of fetal loss (fetal loss between 10 and 21 weeks of gestation)
Fetal death | 5 months
  Rate of fetal death (fetal death from 22 weeks of gestation until delivery)
Neonatal death | 9 months
  Rate of neonatal death (death from birth until 28 days)
Neonatal morbidity | 9 months
  Neonatal morbidity (stay in a neonatal intensive care unit, assisted ventilation > 24 hours, hyaline membrane disease, intraventricular hemorrhages stage III or IV)
Toxicity of aspirin | 8 months
  Potential toxicity of the treatment: major maternal bleeding event (active externalized, intracranial, intra-ocular, retroperitoneal, articular), or minor,
Adherence | 8 months
  Adherence of treatment (diary) and its relationship with the efficacy of the preventive effect on primary outcome,
Biological response to the treatment | 4 months
  Response to the treatment by a urine thromboxane assay
Angiogenic profile | 9 months
  Circulating and urinary angiogenic profile associated with maternal and fetal clinical data: sFLT1 ( Soluble fms-like tyrosine kinase-1)(serum and urine), PlGF ( Placental Growth Factor)(serum and urine)
Child development | 2 years
  Child psychomotor development and health problems at 2 years of age
Child development | 4 years
  Child psychomotor development and health problems at 4 years of age
Subgroups analysis | 9 months
  Rate of the composite morbidity-mortality criterion in 2 subgroups: treatment started before or after 15 SA

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Antoine Béclère, AP-HP, Clamart
  - Hôpital Louis Mourier, AP-HP, Colombes
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU Dijon, Dijon
  - CHU Bicêtre, AP-HP, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - CHU Lyon, Lyon
  - Hôpital St Joseph, Marseille
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Cochin- Port Royal, AP-HP, Paris
  - CHU Robert Débré, AP-HP, Paris
  - CHU Tenon, Paris
  - Hôpital Trousseau, AP-HP, Paris
  - CH Poissy, Poissy
  - CHU St Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No